CLINICAL TRIAL: NCT03928327
Title: A Phase 1 Study of Oral TAK-788 to Evaluate the Drug-Drug Interaction With Itraconazole and Rifampin in Healthy Adult Subjects
Brief Title: A Study to Evaluate Drug-Drug Interaction of TAK-788 With Itraconazole and Rifampin in Healthy Adult Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: TAK-788-1006
Record Dates: First submitted 2019-04-24; First posted 2019-04-26 (Actual); Results first posted 2020-08-21 (Actual); Last update posted 2020-08-21 (Actual); Status verified 2020-08

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — mobocertinib; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1, Treatment Sequence AB (Experimental): TAK-788 20 mg, capsule, at Hour 0 on Day 1 followed by an overnight fast (Treatment A). Following Treatment A, participants received itraconazole 200 mg solution, orally, once daily (QD) on Days 1 to Day 14 and a single oral dose of TAK-788 20 mg capsule was coadministered on Day 5 (Treatment B). There was a washout period of 7 days between the two treatments.
  Interventions: Drug: TAK-788; Drug: Itraconazole
- Part 2, Treatment Sequence CD (Experimental): TAK-788 160 mg, orally, at Hour 0 on Day 1 following an overnight fast (Treatment C). Following Treatment C, participants received rifampin 600 mg as capsules, orally, once daily (QD) on Days 1 to 13 and TAK-788 160 mg as capsules, orally was coadministered on Day 7 (Treatment D). There was a washout period of 7 days between the two treatments.
  Interventions: Drug: TAK-788; Drug: Rifampin

INTERVENTIONS:
Drug: TAK-788 — TAK-788 Capsules
  Other Names: Mobocertinib
Drug: Itraconazole — Itraconazole Oral solution
  Arms: Part 1, Treatment Sequence AB
Drug: Rifampin — Rifampin Capsules
  Arms: Part 2, Treatment Sequence CD

SUMMARY:
The purpose of this study is to characterize the effect of itraconazole (Part 1) and rifampin (Part 2) on the single-dose pharmacokinetics (PK) of TAK-788 and its active metabolites (AP32960 and AP32914) in healthy adult participants.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-788 (Mobocertinib). The study assessed the drug-drug interaction of TAK-788 with either a strong cytochrome P-450 (CYP)3A inhibitor, itraconazole (Part 1) or with a strong CYP3A inducer, rifampin (Part 2) in healthy adult participants.

The study enrolled 24 healthy participants. The study was designed to consist of 2 parts: Part 1- TAK-788 assessment with itraconazole Part 2- TAK-788 assessment with rifampin. Part 1 had 2 cohorts:

Part 1: Participants (n = 12) received a single oral dose of 20 mg capsule of TAK-788 on Day 1 of Period 1 followed by 200 mg itraconazole oral solution once daily (QD) in Period 2 on Days 1 to Day 14 and a single oral dose of TAK-788 20 mg capsule were coadmistered on Day 5 of Period 2.

In Part 2 participants (n = 12) received a single oral 160 mg dose of TAK-788 capsules in Period 1 of Day 1 followed by 600 mg capsules of rifampin QD in Period 2 Days 1 to Day 13 and a single dose of 160 mg TAK-788 capsules was coadministered on Day 7 of Period 1. There was a washout period of 7 days between the dose of TAK-788 on Period 1 and the first dose of rifampin in Period 2.

This single-center trial was conducted in the United States. The overall time to participate in this study was approximately 120 days (including screening period). Participants were contacted by telephone 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Continuous non smoker who has not used nicotine containing products for at least 3 months prior to the first dose and throughout the study based on participant self-reporting.
2. Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs, or electrocardiograms (ECGs), as deemed by the Investigator or designee. Has liver function tests (LFTs) including alanine aminotransferase (ALT), aspartate aminotransferase (AST), alkaline phosphatase (ALP), and total bilirubin within the upper limit of normal at screening and at first check-in.
3. Normal baseline spirometry for forced vital capacity (FVC) and forced expiratory volume (FEV1)/FVC within 7 days prior to the first dosing based on the following normal FVC and FEV1/FVC range: a. 20 - 39 years of age: ≥ 80% and b. 40 - 55 years of age: ≥ 75%
4. Body mass index (BMI) ≥18.0 and ≤32.0 kg/m^2, at screening.

Key Exclusion Criteria:

1. History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing.
2. History or presence of hypersensitivity or idiosyncratic reaction to the study drugs or related compounds.
3. Presence of an acute lung infection, within 3 months of screening.
4. History or presence of any previous lung disease.
5. Part 1 only: History or presence of any of the following, deemed clinically significant by the PI or designee, and as confirmed by the Sponsor:

   * Ventricular dysfunction or risk factors for Torsades de Pointes (e.g., heart failure, cardiomyopathy, family history of Long QT Syndrome);
   * Uncorrected hypokalemia (potassium levels <3.7) and/or hypomagnesemia (magnesium levels <1.9);
   * Myasthenia gravis.
6. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
7. Seated blood pressure is less than 90/40 mmHg or greater than 140/90 mmHg at screening.
8. Seated heart rate is lower than 40 bpm or higher than 99 bpm at screening.
9. QTcF interval is >460 msec (males) or >470 msec (females) or ECG findings are deemed abnormal with clinical significance by the Investigator or designee at screening.
10. Estimated creatinine clearance <90 mL/min at screening
11. Unable to refrain from or anticipates the use of:

    * Any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Medication listed as part of acceptable birth control methods will be allowed. Thyroid hormone replacement medication may be permitted if the subject has been on the same stable dose for the immediate 3 months prior to the first dosing. Acetaminophen (up to 2 g per 24 hour period) may be permitted during the study, only after initial dosing.
    * Any drugs known to be inhibitors or inducers of CYP3A enzymes and/or P-gp, including St. John's Wort, within 28 days prior to the first dosing and throughout the study. Appropriate sources (e.g., Flockhart Table™) will be consulted to confirm lack of pharmacokinetic (PK)/pharmacodynamics interaction with study drugs.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Celerion, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

REFERENCES:
- [Derived] Zhang S, Jin S, Griffin C, Feng Z, Lin J, Venkatakrishnan K, Gupta N. Effects of Itraconazole and Rifampin on the Pharmacokinetics of Mobocertinib (TAK-788), an Oral Epidermal Growth Factor Receptor Inhibitor, in Healthy Volunteers. Clin Pharmacol Drug Dev. 2021 Sep;10(9):1044-1053. doi: 10.1002/cpdd.967. Epub 2021 Jun 19. PMID 34145979

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study in the United States from 02 May 2019 to 16 August 2019.
Pre-assignment Details: Healthy participants were enrolled in this 2-period study to receive: TAK-788 20 mg (Treatment A) along with itraconazole 200 mg (Treatment B) and TAK-788 160 mg (Treatment C) with rifampin 600 mg (Treatment D) in sequential manner to evaluate drug-drug interaction.
Period: Period 1
Arm/Group | Part 1, Treatment Sequence AB | Part 2, Treatment Sequence CD
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period
Arm/Group | Part 1, Treatment Sequence AB | Part 2, Treatment Sequence CD
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Period 2
Arm/Group | Part 1, Treatment Sequence AB | Part 2, Treatment Sequence CD
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Set included participants who received at least one dose of a study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1, Treatment Sequence AB | Part 2, Treatment Sequence CD | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Full Range); unit: years] | 37.7 [26 to 55] | 40.3 [25 to 55] | 39 [26 to 55]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 8 | 4 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 10 | 19
  Not Hispanic or Latino | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 10 | 12 | 22
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 12 | 12 | 24
Weight [Mean (Full Range); unit: Kg] | 85.53 [69.9 to 99.0] | 79.78 [65.1 to 98.9] | 82.65 [65.1 to 99.0]
Height [Mean (Full Range); unit: cm] | 172.8 [157 to 184] | 165.8 [155 to 178] | 169.3 [155 to 184]
Body Mass Index (BMI) [Mean (Full Range); unit: kg/m^2] — Body Mass Index (BMI) was calculated as weight (kg)/[height (m)^2].
  kg/m^2 | 28.573 [25.39 to 31.22] | 28.955 [23.65 to 31.90] | 28.764 [23.39 to 31.90]

OUTCOME MEASURES:

1. Primary Outcome: Treatment B vs Treatment A (Part 1), Combined Molar Exposure for Cmax: Maximum Observed Plasma Concentration of TAK-788, AP32960, and AP32914
Description: The combined molar exposure Cmax for TAK-788 and its metabolites AP32960 and AP3914 value was calculated as the sum of each molar Cmax which was multiplied by 1000 and divided by molecular weight of each analyte, TAK-788, AP32960, and AP32914 respectively. The combined molar exposure was presented in nanomolar.
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: Pharmacokinetic (PK) Set included participants who complied sufficiently with the protocol and display an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Part 1, Treatment A: TAK-788 20 mg, capsule, at Hour 0 on Day 1 followed by an overnight fast in Period 1.
- Part 1, Treatment B: Following Treatment A, participants received itraconazole 200 mg solution, orally, once daily (QD) on Days 1 to Day 14 and a single oral dose of TAK-788 20 mg capsule was coadministered on Day 5 in Period 2.
Arm/Group | Part 1, Treatment A | Part 1, Treatment B
Number analyzed (Participants) | 12 | 12
nM | 13.7 (30.7) | 39.2 (21.1)
Statistical Analysis 1: Comparison: Part 1, Treatment A vs Part 1, Treatment B; Test type: Other; Geometric Least Squares (LS) Mean Ratio = 2.86, 90% CI 2-sided [2.48 to 3.30] — Linear mixed-effects model was used for analysis, using fixed-effect(treatment), random-effect(participants). Geometric mean ratios(GMR), 90% confidence interval(CI) calculated using exponentiation of treatment least squares means(LSMs) difference

2. Primary Outcome: Treatment D Vs Treatment C (Part 2), Combined Molar Exposure for Cmax: Maximum Observed Plasma Concentration of TAK-788, AP32960, and AP32914
Description: as for outcome 1
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: PK Set included participants who complied sufficiently with the protocol and display an evaluable PK profile.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nM
Groups:
- Part 2, Treatment C: TAK-788 160 mg, orally, at Hour 0 on Day 1 following an overnight fast in Period 1.
- Part 2, Treatment D: Following Treatment C, participants received rifampin 600 mg as capsules, orally, once daily (QD) on Days 1 to 13 and TAK-788 160 mg as capsules, orally was coadministered on Day 7 in Period 2.
Arm/Group | Part 2, Treatment C | Part 2, Treatment D
Number analyzed (Participants) | 12 | 12
nM | 177 (34.1) | 14.9 (68.0)
Statistical Analysis 1: Comparison: Part 2, Treatment C vs Part 2, Treatment D; Test type: Other; Geometric LS Mean Ratio = 0.08, 90% CI 2-sided [0.07 to 0.11] — Linear mixed-effects model was used for analysis, using fixed-effect (treatment) and random-effect (participants). GMR and 90% CI was calculated using exponentiation of treatment LSMs difference

3. Primary Outcome: Treatment B Vs Treatment A (Part 1), Combined Molar Exposure for AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration of TAK-788, AP32960, and AP32914
Description: The combined molar exposure AUC∞ for TAK-788 and its metabolites AP32960 and AP3914 value was calculated as the sum of each molar AUC∞ which was multiplied by 1000 and divided by molecular weight of each analyte, TAK-788, AP32960, and AP32914 respectively. The combined molar exposure was presented in hour*nanomolar.
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: PK Set included participants who complied sufficiently with the protocol and display an evaluable PK profile. Overall number analyzed is the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Part 1, Treatment A | Part 1, Treatment B
Number analyzed (Participants) | 8 | 10
hr*nM | 298 (35.2) | 1820 (18.0)
Statistical Analysis 1: Comparison: Part 1, Treatment A vs Part 1, Treatment B; Test type: Other; Geometric LS Mean Ratio = 6.27, 90% CI 2-sided [5.20 to 7.56] — [estimate comment as in outcome 2, analysis 1]

4. Primary Outcome: Treatment D Vs Treatment C (Part 2), Combined Molar Exposure for AUC∞: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration of TAK-788, AP32960, and AP32914
Description: as for outcome 3
Time Frame: Day 1 pre-dose and at multiple time points (up to 168 hours) post-dose
Population: PK Set included participants who complied sufficiently with the protocol and display an evaluable PK profile. Overall number analyzed is the number of participants with data available for analyses. Overall number analyzed is the number of participants with data available for analyses.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*nM
Arm/Group | Part 2, Treatment C | Part 2, Treatment D
Number analyzed (Participants) | 12 | 11
hr*nM | 3610 (43.2) | 194 (70.2)
Statistical Analysis 1: Comparison: Part 2, Treatment C vs Part 2, Treatment D; Test type: Other; Geometric LS Mean Ratio = 0.05, 90% CI 2-sided [0.04 to 0.07] — [estimate comment as in outcome 2, analysis 1]

5. Primary Outcome: Tmax - Time to Reach the Maximum Plasma Concentration (Cmax) of TAK-788
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: PK Set included participants who complied sufficiently with the protocol and display an evaluable PK profile.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1, Treatment A | Part 1, Treatment B | Part 2, Treatment C | Part 2, Treatment D
Number analyzed (Participants) | 12 | 12 | 12 | 12
hr | 6.00 [2.00 to 8.00] | 8.00 [5.99 to 12.00] | 6.00 [4.00 to 8.00] | 4.00 [1.03 to 6.00]

6. Primary Outcome: Tmax - Time to Reach the Maximum Plasma Concentration (Cmax) of AP32960
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: PK Set included participants who complied sufficiently with the protocol and display an evaluable PK profile.
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1, Treatment A | Part 1, Treatment B | Part 2, Treatment C | Part 2, Treatment D
Number analyzed (Participants) | 12 | 12 | 12 | 12
hr | 6.00 [2.00 to 6.01] | 8.00 [6.00 to 12.00] | 6.00 [2.01 to 6.00] | 2.00 [1.03 to 6.00]

7. Primary Outcome: Tmax - Time to Reach the Maximum Plasma Concentration (Cmax) of AP32914
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 3
Measure: Median (Full Range); unit: hr
Arm/Group | Part 1, Treatment A | Part 1, Treatment B | Part 2, Treatment C | Part 2, Treatment D
Number analyzed (Participants) | 9 | 8 | 12 | 8
hr | 6.00 [2.00 to 8.00] | 8.00 [6.00 to 12.00] | 6.00 [4.00 to 6.01] | 4.00 [1.03 to 119.92]

ADVERSE EVENTS:
Time Frame: From first dose up to 30 days post last dose of study drug (Up to 45 days)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Part 1, Treatment A | Part 1, Treatment B | Part 2, Treatment C | Part 2, Treatment D
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 1/12 | 4/12 | 9/12 | 10/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1, Treatment A (N=12) | Part 1, Treatment B (N=12) | Part 2, Treatment C (N=12) | Part 2, Treatment D (N=12)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 2 | 2 | 3
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Oral discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 0 | 2
Chills (General disorders) | 0 | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 1
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 1 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Sensory disturbance (Nervous system disorders) | 0 | 1 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 1
Menstruation delayed (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (2):
  • Study Protocol (2019-04-16): https://cdn.clinicaltrials.gov/large-docs/27/NCT03928327/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-06): https://cdn.clinicaltrials.gov/large-docs/27/NCT03928327/SAP_001.pdf